CLINICAL TRIAL: NCT01296776
Title: Effects of Whole-Body Electromyostimulation on Osteoporosis and Sarcopenia in Independently Living, Frail Elderly Females
Brief Title: Effect of Electromyostimulation on Bone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: City of Erlangen (Unknown); Behinderten- und Versehrten-Sportverband Bayern e.V. (Other); Institute of Physical Education and Sports Sciences (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Professor Dr., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMS-Bone-2011; EK_NO. 4184/2010; EMS_Bone_2011/2012 (Other Grant/Funding Number: IMP_2011)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2012-08

CONDITIONS: Osteopenia; Sarcopenia; Falls
Keywords: exercise; whole-body electromyostimulation; bone mineral density; falls; physical fitness; pain
MeSH Terms: conditions — Bone Diseases, Metabolic; Sarcopenia; Motor Activity; Pain | interventions — Pliability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- whole-body electromyostimulation (Active Comparator): 20 min of whole-body electromyostimulation with sequences of 6 sec of current and 4 sec at 85 Hz performed during low-intensity/low amplitude movements. 3 sessions / 14 days for 12 months
  Interventions: Device: whole-body electromyostimulation
- wellness control group (Placebo Comparator): Low intensity, low frequency exercise that focus on well being. 1 session/week for 10 weeks. 10 blocks of exercise with intermittent periods of 100 weeks of rest
  Interventions: Other: wellness control group.

INTERVENTIONS:
Other: wellness control group. — Light physical exercise and relaxation program once a week in blocks of 10 weeks with breaks of 10 weeks between the blocks. The low-intensity, low-volume program was designed to avoid impact on our endpoints.
  Other Names: functional gymnastic, flexibility, relaxation.
  Arms: wellness control group
Device: whole-body electromyostimulation — 3 sessions of 18 min/14 (1,5 x week)days over 12 months. 10 low-intensity/low amplitude exercises with electromyostimulation equipment with 85 Hz with periods of 6 sec of current and 4 sec of rest.
  Other Names: Electromusclestimulation, electrostimulation; Miha-bodytec
  Arms: whole-body electromyostimulation

SUMMARY:
Although there is some evidence that whole body electromyostimulation(WB-EMS) affect bone via its acute and longitudinal effects on muscle mass and strength, the corresponding impact on bone density and falls in older adults has not been assessed yet. The investigators hypothesize that WB-EMS significantly affects bone parameters as assessed by DXA, and significantly reduce fall rate and ratio in a cohort of frail elderly women.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* 70 years and older
* osteopenia according to WHO
* BMI < 24 kg/m2
* living independently in the area of Erlangen-Nurnberg

Exclusion Criteria:

* medication or diseases affecting bone metabolism (including HRT)
* > 1 hour/week of exercise
* epilepsy, grave neurologic disturbances,
* cardiac pacemaker, grave circulatory disorders,
* abdomen/groin hernia,
* tuberculosis,
* cancer,
* inflammable diseases,
* bleeding tendencies,

Ages: 70 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density at the lumbar spine and femoral neck region | baseline - after 12 months
  Bone Mineral Density as assessed by Dual Energy X-ray Absorptiometry
Falls | throughout the 12 month study period
  Fall frequency and fall related injuries as assessed by the calendar method

SECONDARY OUTCOMES:
maximum strength (trunk and leg extension, grip strength) | baseline - after 12 months
Pain frequency and magnitude at various skeletal sites (including low back pain) | baseline - after 12 months
  as assessed by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Willi A Kalender, PhD, MD, Study Chair — University of Erlangen-Nürnberg Medical School; Wolfgang Kemmler, PhD, Principal Investigator — University of Erlangen-Nürnberg Medical School; Simon von Stengel, PhD, Study Director — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nürnberg, Erlangen, Germany

REFERENCES:
- [Background] Kemmler W, Schliffka R, Mayhew JL, von Stengel S. Effects of whole-body electromyostimulation on resting metabolic rate, body composition, and maximum strength in postmenopausal women: the Training and ElectroStimulation Trial. J Strength Cond Res. 2010 Jul;24(7):1880-7. doi: 10.1519/JSC.0b013e3181ddaeee. PMID 20555279
- [Background] Kemmler W, von Stengel S, Engelke K, Haberle L, Kalender WA. Exercise effects on bone mineral density, falls, coronary risk factors, and health care costs in older women: the randomized controlled senior fitness and prevention (SEFIP) study. Arch Intern Med. 2010 Jan 25;170(2):179-85. doi: 10.1001/archinternmed.2009.499. PMID 20101013
- [Background] von Stengel S, Kemmler W, Engelke K, Kalender WA. Effects of whole body vibration on bone mineral density and falls: results of the randomized controlled ELVIS study with postmenopausal women. Osteoporos Int. 2011 Jan;22(1):317-25. doi: 10.1007/s00198-010-1215-4. Epub 2010 Mar 20. PMID 20306017